CLINICAL TRIAL: NCT04477330
Title: Cortical Priming to Optimize Gait Rehabilitation: Renewal
Brief Title: Cortical Priming to Optimize Gait Rehabilitation in Stroke: a Renewal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: University of Maryland, College Park (Other); Northwestern University (Other)
Responsible Party: Principal Investigator, Sangeetha Madhavan, Professor, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020-0502
Record Dates: First submitted 2020-07-09; First posted 2020-07-20 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: tDCS; Walking
MeSH Terms: conditions — Stroke | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Priming+HIISTT (Experimental): Facilitatory transcranial direct current stimulation (tDCS) and ankle motor training before high intensity interval speed based treadmill training
  Interventions: Other: Transcranial direct current stimulation (tDCS); Other: Ankle motor training; Behavioral: High intensity interval speed based treadmill training (HIISTT)
- Sham+HIISTT (Sham Comparator): Sham tDCS before high intensity interval speed based treadmill training
  Interventions: Behavioral: High intensity interval speed based treadmill training (HIISTT)

INTERVENTIONS:
Other: Transcranial direct current stimulation (tDCS) — 1 mA tDCS
  Arms: Priming+HIISTT
Other: Ankle motor training — Visuomotor target tracking task
  Arms: Priming+HIISTT
Behavioral: High intensity interval speed based treadmill training (HIISTT) — Each treadmill session to include warm-up, high intensity speed-based intervals interleaved with active recovery, and cool down.

SUMMARY:
Achieving functional ambulation post stroke continues to be a challenge for stroke survivors, clinicians, and researchers. In the effort to enhance outcomes of motor training, cortical priming using brain stimulation has emerged as a promising adjuvant to conventional rehabilitation. This project focuses on the development of a long term gait rehabilitation protocol using brain stimulation to improve walking outcomes in people with stroke. The project will also aim to understand the neural mechanisms that are associated with response to the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years
* First ever monohemispheric stroke > 3 months since onset
* Residual hemiparetic gait deficits (e.g. abnormal gait pattern)
* Able to walk for 5 minutes at self-paced speed. Handheld assistive device is acceptable.
* Walking speed lesser than 1.2 m/s
* Lower limb Fugl-Meyer Motor score between 15-30
* At least 5 deg of ankle dorsiflexion necessary to perform the ankle-tracking task

Exclusion Criteria:

* General exclusion criteria

  * Severe osteoporosis
  * Contracture-limiting range of motion of lower limb
  * Score of more than 2 on the Modified Ashworth Scale (indicating increased muscle tone through ankle range of motion)
  * Uncontrolled anti-spasticity medications during the study period
  * Score less than 6 on the Fugl-Meyer Sensory Assessment Scale for the Lower Limb
  * Cardiorespiratory or metabolic diseases (e.g. cardiac arrhythmia, uncontrolled hypertension or diabetes, chronic emphysema)
  * Unhealed decubiti, persistent infection
  * Significant cognitive or communication impairment (Mini-Mental State Examination (MMSE)<21), which could impede the understanding of the purpose of procedures of the study or prevent the patient from performing the ankle-tracking task.
  * Lesions involving the brainstem and cerebellum
  * Failure to pass the graded exercise stress test

TMS exclusion criteria

* Implanted cardiac pacemaker
* Metal implants in the head or face
* Unexplained, recurring headaches
* History of seizures or epilepsy
* Currently under medication that could increase motor excitability and lower seizure threshold
* Skull abnormalities or fractures
* Concussion within the last 6 months
* Currently pregnant

tDCS exclusion criteria

* Skin hypersensitivity
* History of contact dermatitits
* History of allodynia and/or hyperalgesia
* Any other skin or scalp condition that could be aggravated by tDCS

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Walking speed with 10 meter walk test | Change from baseline to immediately after training and baseline to 3 months follow up
  Self-selected and fastest gait speed will be measured as the average of 3 trials of the 10-m walk test (10MWT).

SECONDARY OUTCOMES:
Walking spatiotemporal characteristics with GAITRite walkway | Change from baseline to immediately after training and baseline to 3 months follow up
  Spatiotemporal parameters of walking will be assessed using a 7m long pressure sensitive mat (GAITRite walkway).
Motor impairment with Fugl Meyer Lower Extremity Scale | Change from baseline to immediately after training and baseline to 3 months follow up
  Lower extremity impairment will be measured using the Fugl Meyer Lower Extremity Scale (FMLE), a series of tests of movement, reflex activity, coordination/speed, sensation, and range of motion. The maximum score is 34 and a high score indicates less impairment
Walking endurance with 6-minute walk test | Change from baseline to immediately after training and baseline to 3 months follow up
  Walking endurance will be measured using the 6-Minute Walk test. Participants will walk as far as possible within 6 minutes.
Ankle range of motion | Change from baseline to immediately after training and baseline to 3 months follow up
  Ankle range of motion will be measured using a wireless electrogoniometer affixed to the ankle.
Ankle motor control | Change from baseline to immediately after training and baseline to 3 months follow up
  The participant will track a computer-generated sinusoidal target with ankle dorsiflexion and plantarflexion in a custom-built ankle-tracking device. Accuracy of tracking the target with ankle motion will be calculated.
Balance with mini Balance Evaluations Systems Test (miniBESTest) | Change from baseline to immediately after training and baseline to 3 months follow up.
  Balance will be tested with the Mini-BESTest, involving 14 different tasks to challenge balance.
Aerobic capacity | Change from baseline to immediately after training.
  Cardiopulmonary exercise tests will be performed on a motorized treadmill following an individualized protocol using standard procedures. Measures relating to peak oxygen consumption (VO2 max) will be calculated.
Quality of Life with EuroQol-5D (EQ-5D) | Change from baseline to immediately after training.
  Quality of life will be measured with the EuroQol-5D (EQ-5D), a questionnaire with questions designed to assess aspects of quality of life.
Disability with Modified Rankin Scale | Change from baseline to immediately after training and baseline to 3 months follow up.
  Global disability will be measured with the modified Rankin Scale, a simple 0-6 rating scale.
Community ambulation with wearable sensors | Change from baseline to immediately after training.
  Daily ambulation will be assessed using an accelerometer.
Serum brain derived neurotrophic growth factor (BDNF) | Change from baseline to immediately after training.
  5 ml of blood will be collected from a vein in the participants' arms
Corticomotor excitability using transcranial magnetic stimulation | Change from baseline to immediately after training and baseline to 3 months follow up.
  Corticomotor excitability of the paretic and non-paretic lower limb muscles such as the tibialis anterior and soleus muscle representations will be measured with single pulse transcranial magnetic stimulation (TMS).
Cognitive function using Mini Mental Screening Examination | Change from baseline to immediately after training and baseline to 3 months follow up.
  30-point questionnaire used to capture orientation, attention, memory and language.
Depression using Patient Health Questionnaire-9 (PHQ-9) | Change from baseline to immediately after training and baseline to 3 months follow up.
  The 9-point questionnaire is used to measure degree of depression.
Modified Ashworth Scale | Change from baseline to immediately after training and baseline to 3 months follow up.
  The modified Ashworth scale is a muscle tone assessment scale used to assess the resistance experienced during passive range of motion,

CONTACTS AND LOCATIONS:
Overall Officials: Sangeetha Madhavan, Principal Investigator — University of Illinois at Chicago
Locations (1):
- Physical Therapy, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cleland BT, Madhavan S. The Association of Interlimb Coordination and Temporal Symmetry With Walking Function and Motor Impairment After Stroke. Am J Phys Med Rehabil. 2024 Dec 1;103(12):1104-1109. doi: 10.1097/PHM.0000000000002522. Epub 2024 May 6. PMID 38709654